CLINICAL TRIAL: NCT06372015
Title: Changes in the Lipidomic, Immunological and Circulating microRNA Profile in Patients With Hepatobiliary Pathology, Suffering From Morbid Obesity Undergoing a Dietary Program or Bariatric Surgery
Brief Title: Changes in the Lipidomic, Immunological and miRNA Profile in Patients Undergoing a Dietary Program or Bariatric Surgery
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Collaborators: Notarnicola Maria (Unknown); Cozzolongo Raffaele (Unknown); Shahini Endrit (Unknown); De Pergola Giovanni (Unknown); Lippolis Giuseppe (Unknown)
Responsible Party: Principal Investigator, Dr. Rossella Donghia, Biologyst, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Other Study IDs: RC2023-24
Record Dates: First submitted 2024-04-05; First posted 2024-04-17 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Liver Disease Parenchymal
Keywords: Obesity; Liver Diseases; Bariatric Surgery
MeSH Terms: conditions — Obesity; Liver Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group - Nutritional Approach: Patients who, after a multidisciplinary visit, are found to be ineligible for bariatric surgery.
  Interventions: Other: Nutritional Approach
- Case group - Surgery Approach: Patients who, after a multidisciplinary visit, are referred for bariatric surgery.
  Interventions: Other: Surgery Approach

INTERVENTIONS:
Other: Nutritional Approach — Nutritional Approach
  Groups: Control group - Nutritional Approach
Other: Surgery Approach — Bariatric surgery
  Groups: Case group - Surgery Approach

SUMMARY:
Obesity is a chronic disease characterized phenotypically by an increase in body weight (BMI>30 kg/m2) and by a series of associated pathologies, such as hypertension, diabetes, hepatic steatosis.

The association of these pathologies compromises the patient's survival and quality of life. The multifactorial origin of obesity makes its etiopathology difficult to manage. It is often possible to follow only one therapeutic strategy, especially after the so-called standard treatments, such as dietary intervention and physical activity, have not brought benefit to the patient. In these cases, an appropriate treatment for the patient to enjoy significant weight loss is bariatric surgery.

Bariatric surgery refers to all those interventions aimed at reducing weight in those suffering from obesity, and treating the diseases associated with it.

Among the different types of bariatric surgery, the techniques most used in common clinical practice are intragastric balloons, gastric by pass (RYGB) and sleeve gastrectomy.

The choice of the surgeon, assisted by the multidisciplinary team, is binding in the choice of the type of operation to which the patient will be subjected.

DETAILED DESCRIPTION:
Obesity is a chronic disease characterized phenotypically by an increase in body weight (BMI>30 kg/m2) and by a series of associated pathologies, such as hypertension, diabetes, hepatic steatosis.

The association of these pathologies compromises the patient's survival and quality of life. The multifactorial origin of obesity makes its etiopathology difficult to manage. It is often possible to follow only one therapeutic strategy, especially after the so-called standard treatments, such as dietary intervention and physical activity, have not brought benefit to the patient. In these cases, an appropriate treatment for the patient to enjoy significant weight loss is bariatric surgery.

Bariatric surgery refers to all those interventions aimed at reducing weight in those suffering from obesity, and treating the diseases associated with it.

Among the different types of bariatric surgery, the techniques most used in common clinical practice are intragastric balloons, gastric by pass (RYGB) and sleeve gastrectomy.

In our institution, the diagnostic therapeutic care path for the integrated treatment of obese patients (P.D.T.A) is regulated by DDG n. 528 of 10/27/2022, which indicates the path that the patient must follow if he decides to evaluate a Bariatric Surgery procedure.

In order to proceed with this type of approach, the patient must be followed by a multidisciplinary team (the doctor, the dietician, the psychologist and the kinesiologist) so that the patient can significantly improve his state of health.

The choice of the surgeon, assisted by the multidisciplinary team, is binding in the choice of the type of operation to which the patient will be subjected.

Every patient with obesity associated with hepato-biliary pathologies (hepatic steatosis, gallstones or inflammation of the bile ducts), diagnosed by ultrasound of the complete abdomen and Fibroscan, will be directed towards the procedure most suitable for his health status In the event that the surgeon does not deem it appropriate and safe for the patient, proceed with any bariatric surgery, the guidelines and normal clinical practice ("Diagnostic therapeutic care path for the integrated treatment of the obese patient (P.D.T.A)" of the body - DDG no. 528 of 10/27/2022) provide that the patient is directed to a nutritional approach, through the administration of a diet, always with a multidisciplinary contribution, in which the figure of the psychologist plays great importance, since these patients are often affected by Eating Behavior Disorders (DCA) and have altered eating behavior (hyperphagia, gorging, sweet eating, grazing, snacking).

In obese patients candidates for bariatric surgery, weight loss is only the phenotypic aspect of a metabolic change affecting cellular physiology.

Considering this aspect, lipidomics analysis would be a useful approach to evaluate the composition of fatty acids and membranes of an organism, as well as understanding the alteration of the cellular pathways involved. The measurement of small, dense lipoproteins (sdLDL) will be added to the lipidomic profile, which are more common in some dyslipidemias and can be oxidized more easily than larger LDLs which, oxidized in the cell wall, stimulate the production of cytokines and growth factors, resulting in the recruitment of monocytes.

From a biological point of view, obesity, as well as the alteration of metabolism, involves not only a variation of the lipidomic pattern, but also of the inflammatory pattern, with dysregulation of circulating cytokines and the modification of the expression of circulating microRNAs which emerges from the literature are associated with insulin resistance as well as alterations in glucose homeostasis, and regulators of endocrine function.

Adipose tissue has numerous endocrine functions, capable of stimulating an inflammatory response by regulatory T lymphocytes and macrophages. The activation of these immune cells determines the secretion of pro-inflammatory cytokines, such as TNF, IFN-γ, IL-1β, IL-6, IL-8.

The presence of high levels of pro-inflammatory cytokines in circulation has been observed in obese patients, which can determine the establishment of an inflammatory microenvironment in different body areas. Studies in the literature have shown that weight loss achieved with dietary or surgical therapeutic methods can produce different results in the synthesis of inflammatory mediators. Therefore, future studies are necessary to determine the predictive role of inflammatory mediators in patients undergoing bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients (BMI >30kg/m2) suffering from hepato-biliary pathology diagnosed by Fibroscan
* Adult patients (>18 years).

Exclusion Criteria:

* Patients who are not obese or not affected by hepato-biliary pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients with hepato-biliary pathology, who refer to the nutrition clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Variation of lipidomic parameters | at Baseline and at 1 year
  Variation of lipidomic parameters measured by extraction of fatty acids from red blood cells and run in gas chromatography
The effect of intervention on routine blood chemistry parameters, relating to NAFLD and fibrosis | at Baseline and at 1 year
  Evaluate how bariatric surgery affects routine blood chemistry parameters. The following will be taken into consideration: Blood sugar, Glycated hemoglobin, triglycerides, total cholesterol, HDL and LDL, transaminases, γGT, creatinine, uric acid
Variation in the microRNA profile | at Baseline and at 1 year
  Evaluation of microRNA profile change by real-time PCR

CONTACTS AND LOCATIONS:
Overall Officials: Rossella Donghia, Biologyst, Principal Investigator — Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Locations (1):
- IRCCS "Saverio de Bellis", Castellana Grotte, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bischoff SC, Schweinlin A. Obesity therapy. Clin Nutr ESPEN. 2020 Aug;38:9-18. doi: 10.1016/j.clnesp.2020.04.013. Epub 2020 May 11. PMID 32690184
- [Background] Sasaki A, Nitta H, Otsuka K, Umemura A, Baba S, Obuchi T, Wakabayashi G. Bariatric surgery and non-alcoholic Fatty liver disease: current and potential future treatments. Front Endocrinol (Lausanne). 2014 Oct 27;5:164. doi: 10.3389/fendo.2014.00164. eCollection 2014. PMID 25386164
- [Background] Wolter S, Dupree A, Coelius C, El Gammal A, Kluwe J, Sauer N, Mann O. Influence of Liver Disease on Perioperative Outcome After Bariatric Surgery in a Northern German Cohort. Obes Surg. 2017 Jan;27(1):90-95. doi: 10.1007/s11695-016-2253-6. PMID 27272667
- [Background] Ivanova EA, Myasoedova VA, Melnichenko AA, Grechko AV, Orekhov AN. Small Dense Low-Density Lipoprotein as Biomarker for Atherosclerotic Diseases. Oxid Med Cell Longev. 2017;2017:1273042. doi: 10.1155/2017/1273042. Epub 2017 May 7. PMID 28572872
- [Background] Singh S, Muir AJ, Dieterich DT, Falck-Ytter YT. American Gastroenterological Association Institute Technical Review on the Role of Elastography in Chronic Liver Diseases. Gastroenterology. 2017 May;152(6):1544-1577. doi: 10.1053/j.gastro.2017.03.016. PMID 28442120